CLINICAL TRIAL: NCT05941104
Title: The Effect of Frailty on Blood Biology Indicators, Quality of Life and Survival of Patients With Radical Prostatectomy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Anhui Provincial Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: ShanShan Liu
Record Dates: First submitted 2023-06-16; First posted 2023-07-12 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-06

CONDITIONS: Prostatic Neoplasms; Frailty; Blood Biological Indicators; Quality of Life; Survival
MeSH Terms: conditions — Prostatic Neoplasms; Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Frail group
  Interventions: Other: frailty
- Non-frail group

INTERVENTIONS:
Other: frailty — Frailty is a group of common clinical syndromes in the elderly, characterized by systematic, dynamic and reversible, the core of which is the decline of physiological reserves and the destruction of self-balance.
  Groups: Frail group

SUMMARY:
The goal of this observational study is to evaluate the effect of frailty on blood biology indicators, quality of life and survival of patients with radical prostatectomy.

The main questions it aims to answer are:

1. Evaluate the impact of frailty on the blood biological indicators, quality of life and survival of patients with radical prostatectomy, specifically.
2. Describe the longitudinal changes in the quality of life of patients with radical prostatectomy.

Participants will be divided into frail group or non-frail group based on frailty assessment. Researchers will compare the two groups to see the impact of frailty on the blood biological indicators, quality of life and survival.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with prostate cancer (be diagnosed by relevant imaging examinations or pathology);
2. Radical prostatectomy is planned;
3. Voluntarily sign the informed consent form.

Exclusion Criteria:

1. Diagnosed with other malignant tumors at the same time;
2. Patients with acute infection.

Min Age: 60 Years | Sex: Male
Age Groups: Adult, Older Adult
Study Population: Prostate cancer patients with Radical Prostatectomy.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-07-15 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of Quality of Life from baseline(Quality of Life is a generic concept reflecting concern with the modification and enhancement of life attributes, e.g., physical, political, moral, social environment as well as health and disease.) | baseline(date of hospitalization); 1 month after operation; 3 months after operation; 6 months after operation; 1 year after operation; 2 years after operation.
  Quality of life will be measured by the Extended Prostate Cancer Composite Index Scale (EPIC-26). EPIC-26 is used to assess the functional status of patients with prostate cancer in various domains over the past 4 weeks. Be si de s, EPIC-26 is used to describe the extent of its affects in life of patients with prostate cancer. EPIC-26 contains 26 items in five areas, including urinary incontinence, urinary tract irritation, defecation function, sexual function, and endocrine disorders. Cronbach α coefficient of the scale was 0.854. The overall score is 100 points, and the lower score means better quality of life.

SECONDARY OUTCOMES:
Blood Biology Indicators(including IL-2, IL-6, IL-8,TNF-α, PSA and et al) | baseline(date of hospitalization); 1 month after operation; 3 months after operation; 6 months after operation; 1 year after operation; 2 years after operation.

OTHER OUTCOMES:
Number of Participants Surviving up to 2 years | From date of hospitalization until the date of death from any cause, assessed up to 2 years.

IPD SHARING:
Plan to Share IPD: Undecided